CLINICAL TRIAL: NCT06980909
Title: A Single-dose, Randomized, Open-label, Three-period, Crossover Pharmacokinetic Study of QLC1101 in Healthy Subjects in the Fasting and Fed State
Brief Title: The Food Effect on Pharmacokinetics Study of QLC1101 in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: QLC1101-102
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Effect of Food

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): fasting, high-fat diet, low-fat diet
  Interventions: Drug: QLC1101
- Group B (Experimental): high-fat diet, low-fat diet, fasting
  Interventions: Drug: QLC1101
- Group C (Experimental): low-fat diet , fasting, high-fat diet
  Interventions: Drug: QLC1101

INTERVENTIONS:
Drug: QLC1101 — QLC1101 is an innovative small molecule inhibitor targeting KRAS G12D with independent intellectual property rights developed by Qilu Pharmaceutical Co., Ltd.QLC1101 can prevent GTP/GDP nucleotide exchange and/or the formation of KRAS G12D/GTP/RAF1 complex and inhibit mutant KRAS-dependent signal transduction by specifically binding to the KRAS G12D target, thereby inhibiting the generation of KRAS G12D mutant tumors.
  Arms: Group A
Drug: QLC1101 — QLC1101 is an innovative small molecule inhibitor targeting KRAS G12D with independent intellectual property rights developed by Qilu Pharmaceutical Co., Ltd.QLC1101 can prevent GTP/GDP nucleotide exchange and/or the formation of KRAS G12D/GTP/RAF1 complex and inhibit mutant KRAS-dependent signal transduction by specifically binding to the KRAS G12D target, thereby inhibiting the generation of KRAS G12D mutant tumors
  Arms: Group B
Drug: QLC1101 — QLC1101 is an innovative small molecule inhibitor targeting KRAS G12D with independent intellectual property rights developed by Qilu Pharmaceutical Co., Ltd.QLC1101 can prevent GTP/GDP nucleotide exchange and/or the formation of KRAS G12D/GTP/RAF1 complex and inhibit mutant KRAS-dependent signal transduction by specifically binding to the KRAS G12D target, thereby inhibiting the generation of KRAS G12D mutant tumors.
  Arms: Group C

SUMMARY:
This randomized, open-label, three-period, three-treatment crossover Phase I clinical trial is designed to evaluate the pharmacokinetic profile of QLC1101 capsules administered as a single oral dose under fasting conditions, following a high-fat meal, and following a low-fat meal in healthy adult subjects. The study will further characterize the food effect on QLC1101 pharmacokinetics.

A total of 18 eligible subjects will be enrolled and randomized into three treatment sequences (A, B, C) using a balanced crossover design, with 6 subjects per sequence. The study comprises three treatment periods separated by appropriate washout intervals. In each period, subjects will receive a single dose of QLC1101 under one of three distinct dietary conditions according to their assigned sequence. Following completion of the first treatment period and a washout phase, subjects will crossover to the next dietary condition in the subsequent period, with this process repeating through all three study periods.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects weigh ≥50 kg, female subjects weigh ≥45 kg.
* BMI is within the range of 18.0~28.0 kg/m2 (including the boundary value).

Exclusion Criteria:

* Those who have a history of allergies to drugs, food, pollen, or other clear allergies, or those who are allergic to the experimental drugs and their ingredients;
* Patients with dysphagia or any disease that affects drug absorption, distribution, metabolism and excretion, especially those with a history of gastrointestinal diseases (such as gastric ulcer, gastric bleeding, long-term diarrhea, etc.)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Cmax | 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 144 hours post dose
  Maximum plasma concentration of QLC1101
AUC | 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 144 hours post dose
  Area under the concentration-time curve of QLC1101.
Tmax | 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 144 hours post dose
  Time of maximum observed concentration of QLC1101
t1/2 | 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 144 hours post dose
  Terminal elimination half-life of QLC1101
CL/F | 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 144 hours post dose
  Apparent total clearance of the drug from plasma after oral administration of QLC1101
VZ/F | 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 144 hours post dose
  Apparent volume of distribution after oral administration of QLC1101.